CLINICAL TRIAL: NCT02442869
Title: Developing Adaptive Interventions for Suicidal College Students Seeking Treatment - SMART
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: The Catholic University of America (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 603856; R34MH104714 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-05-13 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Suicide
Keywords: Suicide; College student mental health; CAMS- Collaborative Assessment and Management of Suicidality; SMART -- Sequential Multiple Assignment Randomized Trial; DBT -- Dialectical Behavior Therapy; ATS -- Adaptive Treatment Strategy
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: This study used a Sequential Multiple Assignment Randomized Trial (SMART) design to pilot 4 adaptive treatment strategies (ATSs): ATS1 - Start with Stage 1 CAMS; if responding, end treatment; if not, continue on to Stage 2 CAMS. ATS2 - Start with Stage 1 CAMS; if responding, end treatment; if not, continue on to Stage 2 DBT. ATS3 - Start with Stage 1 TAU; if responding, end treatment; if not, continue on to Stage 2 CAMS. ATS4 - Start with Stage 1 TAU; if responding, end treatment; if not, continue on to Stage 2 DBT.
  For Stage 1, we hypothesized that CAMS would show more improvement on suicide-related variables than TAU and would be more effective with suicidal college students presenting with less complexity at baseline. We did not identify hypotheses for clinical outcome variables in Stage 2 because it was exploratory in nature and focused on the feasibility and acceptability of implementing a SMART design to address suicidal risk in college students.
Who Masked: Outcomes Assessor
Masking Description: The Independent Evaluator was blind to condition assignment when conducting the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1 TAU plus Stage 2 CAMS (Experimental): Treatment as usual [TAU] -- the treatment typically provided by the counselor for 4-8 weeks
  If participant is responding, treatment ends. Participants who don't respond are then re-randomized to
  Collaborative Assessment and Management of Suicidality (CAMS) for 4-16 weeks
  Interventions: Behavioral: Stage 1 Treatment as usual (TAU); Behavioral: Stage 2 CAMS
- Stage 1 TAU plus Stage 2 DBT (Experimental): Treatment as usual [TAU] -- the treatment typically provided by the counselor for 4-8 weeks
  If participant is responding, treatment ends. Participants who don't respond are then re-randomized to
  Dialectical Behavioral Therapy (DBT) for 4-16 weeks
  Interventions: Behavioral: Stage 1 Treatment as usual (TAU); Behavioral: Stage 2 Dialectical Behavioral Therapy (DBT)
- Stage 1 CAMS plus Stage 2 CAMS (Experimental): Collaborative Assessment and Management of Suicidality (CAMS) for 4-8 weeks
  If participant is responding, treatment ends. Participants who don't respond are then re-randomized to
  Additional Collaborative Assessment and Management of Suicidality (CAMS) for 4-16 weeks
  Interventions: Behavioral: Stage 1 CAMS; Behavioral: Stage 2 CAMS
- Stage 1 CAMS plus Stage 2 DBT (Experimental): Collaborative Assessment and Management of Suicidality (CAMS) for 4-8 weeks
  If participant is responding, treatment ends. Participants who don't respond are then re-randomized to
  Dialectical Behavioral Therapy (DBT) for 4-16 weeks
  Interventions: Behavioral: Stage 1 CAMS; Behavioral: Stage 2 Dialectical Behavioral Therapy (DBT)

INTERVENTIONS:
Behavioral: Stage 1 Treatment as usual (TAU) — 4-8 weeks of the treatment typically provided by that counselor with the caveat that neither DBT nor CAMS can be provided.
  Arms: Stage 1 TAU plus Stage 2 CAMS; Stage 1 TAU plus Stage 2 DBT
Behavioral: Stage 1 CAMS — 4-8 weeks of Collaborative Assessment and Management of Suicidality (CAMS)
  Arms: Stage 1 CAMS plus Stage 2 CAMS; Stage 1 CAMS plus Stage 2 DBT
Behavioral: Stage 2 CAMS — 4-16 weeks of Collaborative Assessment and Management of Suicidality (CAMS)
  Arms: Stage 1 CAMS plus Stage 2 CAMS; Stage 1 TAU plus Stage 2 CAMS
Behavioral: Stage 2 Dialectical Behavioral Therapy (DBT) — 4-16 weeks of Dialectical Behavioral Therapy (DBT)
  Arms: Stage 1 CAMS plus Stage 2 DBT; Stage 1 TAU plus Stage 2 DBT

SUMMARY:
This pilot study tested the feasibility of utilizing an adaptive intervention strategy for college students who are suicidal when first seeking treatment at a campus clinic. Right now, the typical strategy may rely on a "one size fits all" approach, but in fact suicidal students vary greatly on what and how much they need. This study will pave the way for subsequent larger trials for clinical decision making (trying one approach, and if that doesn't work, another) to be empirically developed and tested in a subsequent large-scale multisite trial with the goal of maximizing resources in overburdened college counseling centers. This pilot study followed by a subsequent large-scale trial could eventually significantly impact service delivery to suicidal college students at college counseling centers.

DETAILED DESCRIPTION:
The primary aim of this proposal was to conduct feasibility research to inform the implementation of a future full-scale SMART (sequential, multiple assignment, randomized trial, Almirall et al., 2012) that will be used to construct adaptive treatment strategies (ATSs) to address suicidality in college students seeking services at college counseling centers (CCCs). ATSs individualize treatment via decision rules that can specify how the type and intensity of an intervention should be sequenced based on variables collected mid-treatment (or at baseline), such as response to treatment. Suicidality is a frequent presenting concern among college students seeking treatment; yet, studies with this population show that some students respond rapidly to treatment whereas others may require considerably more resources. However, at this time, CCCs, which are overburdened and often have to resort to waitlists, have no guidance as to how to sequence different approaches with suicidal students in an empirically-based and cost effective manner. Therefore, empirically validated ATSs are needed in the provision of services to suicidal college students to address the heterogeneity of students with this presentation and the variability in response to interventions. In the present pilot SMART, each participant progressed through two stages of intervention. In the first stage (S1) 62 participants were randomized to one of two brief individual therapy interventions for 4-8 weeks: 1) one that is suicidality-focused (Collaborative Assessment and Management of Suicidality (CAMS; Jobes, 2016) and 2) one that relies on Treatment as Usual (TAU) being provided at a CCC. Responders to either program will discontinue services/ be stepped down and be monitored over time for maintenance. Non-responders to either intervention who remain in treatment (estimated n = 18) were re-randomized to one of two second-stage (S2) higher intensity/dosage intervention options for an additional 4-16 weeks: 1) CAMS (either continued but for a longer period of time or administered for the first time) or 2) Comprehensive Dialectical Behavior Therapy (DBT, Linehan, 1993a, 1993b) which includes individual therapy, skills groups, and phone coaching for the clients and DBT peer consultation for the therapists. This study enrolled moderately to severely suicidal (endorsing thoughts of wanting to die of 2 or above on 0-4 scale) college students in the "emerging adulthood" phase (18-25 years of age) seeking services at a CCC. The aims of this feasibility services research project were to 1) develop and refine a SMART design in a CCC setting; 2) assess the feasibility of conducting a SMART and its embedded ATSs in a CCC setting; 3) obtain estimates of overall response rates to S1 interventions; and 4) explore the utility of incorporating secondary tailoring variables (e.g., level of functioning at pre-treatment, ratio of Wish to Live vs. Wish to Die) in the ATSs in the subsequent larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled student at the University of Nevada, Reno (UNR)
* Seeking services at Counseling Services at UNR
* 18 to 25 years of age
* Moderate to severe suicidality (indicated by a score of 2 or above (range is 0 "not at all like me" to 4 "extremely like me") on the Counseling Center Assessment of Psychological Symptoms (CCAPS-34; Locke et al., 2012) question, "I have thoughts of ending my life."

Exclusion Criteria:

* Individual is deemed inappropriate to receive services at UNR Counseling Services by the intake worker (the primary exclusion criterion).
* Participant cannot have been in treatment at UNR Counseling Services within the previous 3 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pistorello, PhD, Principal Investigator — University of Nevada, Reno
Locations (1):
- Counseling Services, University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
After study is complete and data analyzed, interested researchers can contact the PI for data inquiries. Only de-identified data will be released to qualified researchers.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: July 2018 to July 2022
Access Criteria: 1. Researcher contacts PI at pistorel@unr.edu
  2. There is justification for the use of the data and this is deemed appropriate by the PI and institution representative
URL: https://scholarworks.unr.edu/

REFERENCES:
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Almirall D, Compton SN, Gunlicks-Stoessel M, Duan N, Murphy SA. Designing a pilot sequential multiple assignment randomized trial for developing an adaptive treatment strategy. Stat Med. 2012 Jul 30;31(17):1887-902. doi: 10.1002/sim.4512. Epub 2012 Mar 22. PMID 22438190
- [Background] American College Health Association (ACHA, 2012). ACHA-National College Health Assessment II: Reference group executive summary Spring 2011. Hanover MD: American College Health Association.
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] Comtois KA, Jobes DA, S O'Connor S, Atkins DC, Janis K, E Chessen C, Landes SJ, Holen A, Yuodelis-Flores C. Collaborative assessment and management of suicidality (CAMS): feasibility trial for next-day appointment services. Depress Anxiety. 2011 Nov;28(11):963-72. doi: 10.1002/da.20895. Epub 2011 Sep 21. PMID 21948348
- [Background] Center for Collegiate Mental Health (CCMH, 2012). CCAPS 2012 Technical Manual. University Park, PA.
- [Background] Jobes, D. A. (2006). Managing suicidal risk: A collaborative approach. New York: The Guilford Press.
- [Background] Linehan, M.M. (1993). Cognitive behavioral therapy of borderline personality disorder. New York: Guilford Press.
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Linehan, M.M. (2015). DBT skills training manual (2nd ed.). New York, NY: Guilford Press.
- [Result] Pistorello J, Jobes DA, Gallop R, Compton SN, Locey NS, Au JS, Noose SK, Walloch JC, Johnson J, Young M, Dickens Y, Chatham P, Jeffcoat T. A Randomized Controlled Trial of the Collaborative Assessment and Management of Suicidality (CAMS) Versus Treatment as Usual (TAU) for Suicidal College Students. Arch Suicide Res. 2021 Oct-Dec;25(4):765-789. doi: 10.1080/13811118.2020.1749742. Epub 2020 Apr 10. PMID 32275480
- [Result] Pistorello J, Jobes DA, Compton SN, Locey NS, Walloch JC, Gallop R, Au JS, Noose SK, Young M, Johnson J, Dickens Y, Chatham P, Jeffcoat T, Dalto G, Goswami S. Developing Adaptive Treatment Strategies to Address Suicidal Risk in College Students: A Pilot Sequential, Multiple Assignment, Randomized Trial (SMART). Arch Suicide Res. 2017 Oct-Dec;22(4):644-664. doi: 10.1080/13811118.2017.1392915. Epub 2018 Feb 12. PMID 29220633

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 TAU (Participant Responding to Treatment): Treatment as usual [TAU] -- the treatment typically provided by the counselor for 4-8 weeks.
  After 8 weeks or after participants completed their Stage 1 TAU treatment, whichever was later, they returned for their post Stage 1 assessment.
- Stage 1 CAMS (Participant Responding to Treatment): Collaborative Assessment and Management of Suicidality [CAMs] -- treatment provided by counselor for 4-8 weeks.
  After 8 weeks or after participants completed their Stage 1 CAMS treatment, whichever was later, they returned for their post Stage 1 assessment.
- Stage 2 CAMS (Didn't Respond to Stage 1 TAU); Stage 2 CAMS (Didn't Respond to Stage 1 CAMS): Collaborative Assessment and Management of Suicidality (CAMS) -- treatment provided by counselor for 4-16 weeks.
  16 weeks after participants completed their post Stage 1 assessment or after participants completed their Stage 2 CAMS treatment, whichever was later, they returned for their post Stage 2 assessment.
- Stage 2 DBT (Didn't Respond to Stage 1 TAU); Stage 2 DBT (Didn't Respond to Stage 1 CAMS): Dialectical Behavioral Therapy (DBT) course -- treatment provided by counselor for 4-16 weeks.
  16 weeks after participants completed their post Stage 1 assessment or after participants completed their Stage 2 DBT treatment, whichever was later, they returned for their post Stage 2 assessment.
Period: Overall Study
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Started | 18 | 29 | 6 | 2 | 5 | 2
Completed | 13 | 20 | 6 | 1 | 3 | 2
Not Completed | 5 | 9 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage 1 TAU (Participant Responding to Treatment): Treatment as usual (TAU): 4-8 weeks of treatment typically provided by that counselor with the caveat that neither DBT nor CAMS can be provided.
  Participant responded to TAU, treatment ended.
- Stage 1 CAMS (Participant Responding to Treatment): Stage 1 CAMS: 4-8 weeks of Collaborative Assessment and Management of Suicidality (CAMS).
  Participant responded to CAMS, treatment ended.
- Stage 2 CAMS (Didn't Respond to Stage 1 TAU): Participant didn't respond to Stage 1 TAU and was re-randomized to:
  Stage 2 CAMS: 4-16 weeks of Collaborative Assessment and Management of Suicidality (CAMS)
- Stage 2 CAMS (Didn't Respond to Stage 1 CAMS): Participant didn't respond to Stage 1 CAMS treatment and was re-randomized to:
  Stage 2 CAMS: 4-16 additional weeks of Collaborative Assessment and Management of Suicidality (CAMS)
- Stage 2 DBT (Didn't Respond to Stage 1 TAU): Participant didn't respond to Stage 1 TAU treatment and was re-randomized to:
  Dialectical Behavioral Therapy (DBT): 4-16 weeks of Dialectical Behavioral Therapy (DBT)
- Stage 2 DBT (Didn't Respond to Stage 1 CAMS): Participant didn't respond to Stage 1 CAMS treatment and was re-randomized to:
  Dialectical Behavioral Therapy (DBT): 4-16 weeks of Dialectical Behavioral Therapy (DBT)
- Total: Total of all reporting groups
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS) | Total
Number analyzed (Participants) | 18 | 29 | 6 | 2 | 5 | 2 | 62
Age, Continuous [Mean (Full Range); unit: years] | 20.50 [18 to 25] | 19.62 [18 to 24] | 20.50 [18 to 23] | 18.5 [18 to 19] | 20.60 [18 to 24] | 18.50 [18 to 19] | 19.97 [18 to 25]
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 29 | 6 | 2 | 5 | 2 | 62
  > 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 18 | 5 | 1 | 4 | 2 | 42
  Male | 6 | 10 | 1 | 1 | 1 | 0 | 19
  Transgender | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 5 | 0 | 1 | 1 | 0 | 10
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Hispanic/Latino | 1 | 3 | 1 | 0 | 0 | 0 | 5
  White | 6 | 15 | 5 | 1 | 3 | 0 | 30
  More than one race | 8 | 5 | 0 | 0 | 1 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 18 | 29 | 6 | 2 | 5 | 2 | 62

OUTCOME MEASURES:

1. Primary Outcome: Feasibility/Acceptability: Participation Rate
Description: Number of students approached who agreed to participate in the study
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Agreed to Participate: Number of eligible students approached who agreed to participate
- Declined to Participate: Number of eligible students approached who declined to participate
Arm/Group | Agreed to Participate | Declined to Participate
Number analyzed (Participants) | 62 | 30
Participants | 18 | 29

2. Primary Outcome: Feasibility/Acceptability: Number of Students Who Declined to Participate in the Study and Why
Description: Two typologies as to when students declined to participate emerged: Declined when approached, and Declined during the consenting process.
Time Frame: Baseline
Population: Note the 'Overall Number of Participants Analyzed' in this context is the total number of eligible students and not the total number who consented to participate (intent to treat).
Measure: Number; unit: students
Groups:
- Num. of Students Declining & Agreeing to Participate: Number of students who declined to participate in the study and why. Reasons eligible students declined participation in the study are detailed in the Pistorello et al., 2017 publication.
Arm/Group | Num. of Students Declining & Agreeing to Participate
Number analyzed (Participants) | 92
students
  Declined when approached by counselor | 23
  Declined during the consenting process | 7
  Agreed: Enrolled & Randomized in study | 62

3. Primary Outcome: Feasibility/Acceptability: Number of Students Who Were Retained Within Each of the Four Adaptive Treatment Strategies
Description: Feasibility/Acceptability (Treatment Retention): Number of students who were retained within each of the four Adaptive Treatment Strategies
Time Frame: After Stage 2
Population: All participants were assessed at the end of the Stage 2 (approximately 6 months after baseline), regardless of whether they continued into Stage 2 treatments or not
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 18 | 29 | 6 | 2 | 5 | 2
Participants
  Retained | 13 | 20 | 6 | 1 | 3 | 2
  Dropped | 5 | 9 | 0 | 1 | 2 | 0

4. Primary Outcome: Feasibility/Acceptability: General Time to Drop-out Among Students Who Dropped Out Within Each Arm
Description: General time to drop out among students who dropped out within each arm, by number of treatment sessions received
Time Frame: Throughout the 24 weeks of treatment delivery (Stage 1 and Stage 2)
Population: Columns/Arms with zero (0) participants indicates that no participants dropped out of that particular Arm of the study, but note the small sample size.
  All participants were assessed at the end of the Stage 2 (approximately 6 months after baseline), regardless of whether they continued into Stage 2 treatments or not
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 5 | 9 | 0 | 1 | 2 | 0
Participants
  Attended 0 sessions | 0 | 2 | 0 | 0 | 0 | 0
  Attended 1-2 sessions | 2 | 4 | 0 | 0 | 0 | 0
  Attended 3-5 sessions | 1 | 0 | 0 | 0 | 0 | 0
  Attended 6 or more sessions | 2 | 3 | 0 | 1 | 2 | 0

5. Primary Outcome: Feasibility/Acceptability: Fidelity of the CAMS Intervention Delivery by "Real World" CCC Counselors Via the CAMS Rating Scale 3 (CRS.3)
Description: CAMS adherence ratings conducted by CAMS experts. The CAMS Rating Scale (CRS.3) was used to assess CAMS adherence. The CRS.3 has 14 items rated on a 7-point scale from 0 (Poor) to 6 (Excellent). Therefore, higher scores indicate better adherence. Adherence covers various domains: collaboration (4 items), suicide focus (1 item), risk assessment (1 item), treatment planning (3 items), intervention (2 items), and overall adherence (1 item). Two coders assessed the fidelity of CAMS by observing digitally recorded sessions.
Time Frame: Throughout the 24 weeks of treatment delivery (Stage 1 and Stage 2)
Population: The first four sessions of randomly selected CAMS Stage 1 cases were rated for adherence for each counselor. An overall mean and then an overall count of 'Adherent' or 'Not Adherent' was created. The following reported data only reflects the overall adherence ratings (1 item).
  All participants were assessed at the end of the Stage 2 (approximately 6 months after baseline), regardless of whether they continued into Stage 2 treatments or not
Measure: Count of Units; unit: Number of sessions rated for adherence
Units Other Than Participants: Number of sessions rated for adherence
Arm/Group | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 21 | 4 | 2
Number analyzed (Number of sessions rated for adherence) | 50 | 6 | 2
Number of sessions rated for adherence
  # Not Adherent (< 3) | 2 | 0 | 0
  # Adherent (3 or above) | 48 | 6 | 2

6. Primary Outcome: Feasibility/Acceptability: Fidelity of the DBT Intervention Delivery by "Real World" CCC Counselors Via the University of Washington DBT Adherence Rating Scale (Linehan & Korslund, 2003)
Description: DBT adherence ratings conducted by DBT adherence experts. The University of Washington Dialectical Behavior Therapy Adherence Coding Scale (DBTACS) was utilized to check DBT adherence. The DBTACS has various dimensions, each measured on a 5-point scale (ranging from 0.0-5.0, with 5 indicating greater adherence). Therefore, higher scores indicate better adherence. The overall score is an average of these dimensions with a cutoff of 4.0 for adherence.
Time Frame: During Stage 2 (sessions 9 through 24 of treatment)
Population: Approximately 1-2 DBT session tapes per five counselors (two counselors did not have available tapes) were semi-randomly selected and rated for adherence. It should be noted that DBTACS adherence scores are specific to a given session and only when multiple consecutive sessions are rated is the conclusion that a therapist is "adherent" warranted.
Measure: Count of Units; unit: Number of sessions rated for adherence
Units Other Than Participants: Number of sessions rated for adherence
Arm/Group | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 3 | 2
Number analyzed (Number of sessions rated for adherence) | 4 | 3
Number of sessions rated for adherence
  # Not Adherent (Below 4.0) | 0 | 1
  # Adherent (4.0 or above) | 4 | 2

7. Primary Outcome: Feasibility/Acceptability: Satisfaction With Treatment as Reported by Student Participants Via the the Client Satisfaction Questionnaire (CSQ-8)
Description: The Client Satisfaction Questionnaire (CSQ-8) assesses client satisfaction with treatment on a scale from 8-32, with higher scores indicating greater satisfaction. Low satisfaction ratings (CSQ score of 8-20); Medium satisfaction ratings (CSQ score of 21-26); High satisfaction ratings (CSQ score of 27-32).
Time Frame: End of Stage 1 (after 8 weeks of treatment) and end of Stage 2 (after 24 weeks of treatment)
Population: Not all participants completed measures following Stage 2, therefore although fourteen clients were re-randomized to S2, only eleven completed the CSQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 13 | 24 | 5 | 2 | 5 | 2
score on a scale
  Stage 1 | 27.54 (3.99) | 27.96 (4.09) | 27.00 (4.00) | 27.00 (2.82) | 25.00 (2.65) | 28.00 (4.24)
  Stage 2: number analyzed (Participants) | 12 | 23 | 5 | 2 | 3 | 2
  Stage 2 | 27.17 (4.28) | 28.04 (3.64) | 28.80 (3.83) | 22.00 (8.49) | 25.00 (2.00) | 32.00 (0.00)

8. Primary Outcome: Feasibility/Acceptability: Satisfaction With Treatment by Counselors Via the CSQ-8 (Therapist Version)
Description: The Client Satisfaction Questionnaire (CSQ-8) Therapist Version assesses therapist satisfaction with treatment on a scale from 8-32, with higher scores indicating greater satisfaction. Low satisfaction ratings (CSQT score of 8-20); Medium satisfaction ratings (CSQT score of 21-26); High satisfaction ratings (CSQT score of 27-32).
Time Frame: End of Stage 1 (after 8 weeks of treatment) and end of Stage 2 (after 24 weeks of treatment)
Population: The unit of analysis is participants, however, counselors completed the Client Satisfaction Questionnaire Therapist Version (CSQT-8).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
Number analyzed (Participants) | 18 | 28 | 5 | 2 | 5 | 2
score on a scale
  Stage 1 | 26.83 (4.38) | 25.18 (6.51) | 23.33 (5.39) | 21.50 (2.12) | 21.80 (4.60) | 22.00 (2.83)
  Stage 2: number analyzed (Participants) | 17 | 25 | 4 | 2 | 4 | 1
  Stage 2 | 24.59 (6.00) | 25.00 (6.40) | 25.25 (2.50) | 23.00 (5.66) | 23.50 (3.11) | 30.00 (NA) — sample of 1, no Std Dev. to calculate

9. Secondary Outcome: Scale for Suicide Ideation-Current (SSI)
Description: The SSI is an interviewer-rated measure based on 19 questions related to the highest intensity of suicidal ideation in the past 2 weeks, including attitudes, behaviors, and plans. Each item is rated as 0,1, or 2 and the total scale yields a score of 0-38. Higher scores indicate greater suicide risk.
Time Frame: End of Stage 1 interventions - ~8 weeks after baseline; End of Stage 2 interventions ~24 weeks after baseline; and Follow-up (3 months after all treatment has ended) ~36 weeks after baseline
Population: Not all participants were assessed at S1 due to several participants declining assessments or missing the assessment window. Data are only included for S1 treatment arms in line with our pre-specified research aim to obtain estimates of overall response rates to S1 interventions. Clinical outcome variables were not interpreted at Stage 2 because it was exploratory in nature focusing on the feasibility/acceptability of implementing a SMART design to address suicidal risk in college students.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stage 1 TAU: Treatment as usual (TAU): 4-8 weeks of treatment typically provided by that counselor with the caveat that neither DBT nor CAMS can be provided.
Arm/Group | Stage 1 TAU | Stage 1 CAMS
Number analyzed (Participants) | 29 | 33
score on a scale
  Baseline | 13.72 (7.07) | 13.79 (5.13)
  S1 (end of Phase I interventions) -8 weeks: number analyzed (Participants) | 21 | 30
  S1 (end of Phase I interventions) -8 weeks | 7.35 (6.45) | 5.66 (6.44)
Statistical Analysis 1: Comparison: Stage 1 TAU vs Stage 1 CAMS; Due to the large number of zeroes in the Suicidal Ideation (SI)-Current Subscale of the SSI at post (over a third of the participants reported no SI at the end of treatment), a zero-altered model was utilized which divided the outcome into (1) the probability of any SI and (2) the intensity of SI when non-zero, as done in other studies. This analysis tested the difference between the CAMS and TAU arms based on number of participants reporting no SI post Stage 1 treatment; Test type: Superiority; p = 0.19, Chi-squared; Df (1); Net difference in proportion = 1.73, 95% CI 2-sided [-2.41 to 15.35] — NNT = 5.59

10. Other Pre Specified Outcome: The Suicide Attempt and Self-Injury Count (SASI-C)
Description: The SASI-C is a very brief interview of past self-inflicted injuries, categorized into suicide attempts and nonsuicidal acts. The SASI-C creates counts of self-inflicted injuries by method, medical risk severity, and lethality.
Time Frame: The time frame at pretreatment was both lifetime and past 2 months at baseline: and all other assessments focused on the last 2 months. This was assessed at baseline and after Stage 1 (~ 8 weeks later).
Population: Note. Some attrition/respondent drop-out is present throughout this study. Data are only included for S1 treatment arms in line with our pre-specified research aim to obtain estimates of overall response rates to S1 interventions. Clinical outcome variables were not interpreted at Stage 2 because it was exploratory in nature focusing on the feasibility/acceptability of implementing a SMART design to address suicidal risk in college students.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 TAU | Stage 1 CAMS
Number analyzed (Participants) | 29 | 33
Participants
  Baseline : SASI-C (endorsed suicide attempt in last 2 month) | 7 | 3
  Baseline : SASI-C (1 or more self-inflicted injuries) | 24 | 26
  Post Stage 1 : SASI-C (endorsed suicide attempt in last 2 months): number analyzed (Participants) | 23 | 29
  Post Stage 1 : SASI-C (endorsed suicide attempt in last 2 months) | 0 | 0
  Post Stage 1 : SASI-C (1 or more self-inflicted injuries): number analyzed (Participants) | 23 | 29
  Post Stage 1 : SASI-C (1 or more self-inflicted injuries) | 9 | 7
Statistical Analysis 1: Comparison: Stage 1 TAU vs Stage 1 CAMS; Test type: Superiority; p = 0.25, Regression, Logistic; Net difference in proportion = 1.30

11. Other Pre Specified Outcome: The Counseling Center Assessment of Psychological Symptoms (CCAPS-34) Depression Scale.
Description: The CCAPS-34 is a measure of psychological distress with several sub-scales (Depression) specifically designed for college students seeking services. Depression subscale scores range from 0.1-5.0 with lower scores representing less depression
Time Frame: Baseline and End of Stage 1 interventions - 8 weeks after baseline
Population: Note: Some attrition/respondent drop-out is present throughout this study. Data are only included for S1 treatment arms in line with our pre-specified research aim to obtain estimates of overall response rates to S1 interventions. Clinical outcome variables were not interpreted at Stage 2 because it was exploratory in nature focusing on the feasibility/acceptability of implementing a SMART design to address suicidal risk in college students.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 TAU | Stage 1 CAMS
Number analyzed (Participants) | 29 | 33
score on a scale
  Baseline | 1.98 (1.06) | 2.23 (0.99)
  Stage 1: number analyzed (Participants) | 21 | 30
  Stage 1 | 1.70 (0.90) | 1.42 (1.70)
Statistical Analysis 1: Comparison: Stage 1 TAU vs Stage 1 CAMS; Test type: Superiority — Power analyses. We determined that with a sample size of 62 clients, the outcome analyses had at least 80% power to detect an effect size of 0.80 (Ahn etal., 2001); p = 0.035, t-test, 2 sided; t(60) = 2.15; Mean Difference (Net) = 0.55, 95% CI 2-sided [0.04 to 1.05]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during both Phases of the study through the follow-up assessment (approximately 6 months after baseline, for a total of approximately 6 months).
Description: Adverse events were tracked using seven typologies: Death by Suicide, Other Death, Attempted Suicide, Non-Suicidal Self-Injury, Psychiatric Admission, Medical Hospitalization, & Other Serious Adverse Event.
Arm/Group | Stage 1 TAU (Participant Responding to Treatment) | Stage 1 CAMS (Participant Responding to Treatment) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/29 | 0/6 | 0/2 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/6 | 2/2 | 2/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/6 | 0/2 | 0/5 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 TAU (Participant Responding to Treatment) (N=18) | Stage 1 CAMS (Participant Responding to Treatment) (N=29) | Stage 2 CAMS (Didn't Respond to Stage 1 TAU) (N=6) | Stage 2 CAMS (Didn't Respond to Stage 1 CAMS) (N=2) | Stage 2 DBT (Didn't Respond to Stage 1 TAU) (N=5) | Stage 2 DBT (Didn't Respond to Stage 1 CAMS) (N=2)
Death by Suicide (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other Death (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — All mortality other than suicide
Attempted Suicide (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Self-reported by client
Non-Suicidal Self-Injury (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Self-reported by client
Psychiatric Admission (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical Hospitalization (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other Serious Adverse Event (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Client experienced a silent seizure while in treatment.

LIMITATIONS AND CAVEATS:
The study focused on acceptability and feasibility. Although data was collected for Stage 2 and analyzed for acceptability and feasibility outcomes (e.g., CSQ), clinical outcomes (e.g., SSI, CCAPS) were only interpreted for Stage 1 due to small sample sizes among the Stage 2 groups. A larger study is needed to identify the most effective sequence of care for suicidal risk treatments at college counseling centers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No